CLINICAL TRIAL: NCT00256880
Title: A Phase II, Open-Label Study of Pazopanib (GW786034) in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Pazopanib (GW786034) In Subjects With Relapsed Or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEG20006
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Carcinoma, Renal Cell
Keywords: Pazopanib(GW786034); Solid Tumors; Myeloma
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms, Plasma Cell | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW786034

SUMMARY:
The purpose of this study is to determine how effective and safe a new investigational drug is in treating patients with relapsed or refractory multiple myeloma. The treatment involves daily dosing. A patient may continue to receive the treatment as long as they are benefiting from the treatment. Blood samples will be taken at specific times to measure the amount of drug in your body at specific times after the drug is given. Blood samples will also be taken for lab tests such as complete blood counts and clinical chemistries. Physical exams will be performed before each treatment. During the treatment phase, the patients will undergo regular assessments for safety and clinical response.

ELIGIBILITY:
Inclusion criteria:

* Must have diagnosis of relapsed or refractory multiple.
* bone marrow function [ANC (absolute neutrophil count) greater than 1000/mm3]; platelet count greater than or equal to 75,000/mm3.
* renal function (calculated creatinine clearance >50 mL.min, albumin less than or equal to 500 mg).

Exclusion criteria:

* Failed more than 3 prior lines of therapy including stem cell transplant.
* Females who are pregnant or nursing.
* Unstable blood pressure.
* Significant heart conditions or history of thrombosis.
* Any unstable, pre-existing major medical condition or history of other cancers.
* Have received an investigational drug, chemotherapy, radiation treatment or surgery within 28 days prior to entering the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-01; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of GW786034 in patients with relapsed or refractory multiple myeloma (MM).

SECONDARY OUTCOMES:
Evaluate time-to-tumor progression (TTP), time to response, and duration of response. Characterize the pharmacokinetics of GW786034 in patients with MM.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (5):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Seattle, Washington
- Australia (2):
  - GSK Investigational Site, East Melbourne, Victoria
  - GSK Investigational Site, Melbourne, Victoria

REFERENCES:
- [Background] Prince HM, Honemann D, Spencer A, Rizzieri DA, Stadtmauer EA, Roberts AW, Bahlis N, Tricot G, Bell B, Demarini DJ, Benjamin Suttle A, Baker KL, Pandite LN. Vascular endothelial growth factor inhibition is not an effective therapeutic strategy for relapsed or refractory multiple myeloma: a phase 2 study of pazopanib (GW786034). Blood. 2009 May 7;113(19):4819-20. doi: 10.1182/blood-2009-02-207209. No abstract available. PMID 19423744